CLINICAL TRIAL: NCT01641497
Title: Phase III Study Comparing 3D Conformal Radiotherapy and Conformal Radiotherapy IMRT to Treat Endometrial Cancer of 70 Years Old Women : Contribution of Oncogeriatric Evaluation to the Study of Acute Toxicity
Brief Title: Phase III Study Comparing 3D Conformal Radiotherapy and Conformal Radiotherapy IMRT to Treat Endometrial Cancer
Acronym: TOMOGYN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TOMOGYN - 1105; 2011-A01543-38 (Other: DEDIM (ANSM))
Record Dates: First submitted 2012-07-09; First posted 2012-07-16 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; IMRT; age over 70
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D conformational radiotherapy (Active Comparator): 25 * 1.8 Gy in 5 weeks (=45 Gy). 3D conformational radiation
  Interventions: Radiation: 3D conformational radiation
- Intensity-Modulated Radiation Therapy (Experimental): 25 * 1.8 Gy in 5 weeks (=45 Gy). IMRT
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: 3D conformational radiation — 25 * 1.8 Gy in 5 weeks (=45 Gy)
  Arms: 3D conformational radiotherapy
Radiation: IMRT — 25 * 1.8 Gy in 5 weeks (=45 Gy)
  Arms: Intensity-Modulated Radiation Therapy

SUMMARY:
Comparison of radiotherapy tolerance (two types of radiotherapy) for patients over 70 years with a endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer is the most common form of gynecological cancer in France with 6560 new cases in 2010. Endometrial cancers occurs generally after menopause but are sometimes diagnosticated before 40 years. The 5 years Overall survival of endometrial cancer is 76% (95% for non locally advanced or non metastatic disease).

Some factors are involved in disease prognostic: age, geographical origin, physical status, tumor grade, tumor histology and probably biomarkers. Some studies demonstrated that advanced age is a negative prognostic factor due to higher relapse risk and higher specific mortality. Unfortunately, Incidence of endometrial cancer will probably increase in future due to aging of the occidental population.

Current treatment of endometrial cancer is based on post-operative radiation therapy: adjuvant brachytherapy or adjuvant external beam radiation therapy. However these techniques lead to serious toxicity (digestive toxicity, ileitis...) in elder patient. Consequently, pelvic radiation therapy is difficult to organize before 75 years and dangerous to perform after 80 years.

However a new technique called: Intensity-modulated radiation therapy (IMRT) can make the difference. IMRT is a new high precision radiotherapy technique probably well adapted for old people, with less toxicity than current radiotherapy.

Nevertheless, IMRT is not recognized as a standard radiation therapy procedure in France and Europe.

Thus, goal of TOMOGYN study is to compare the tolerance of old women (at least 70 years), with endometrial cancer, treated with external beam radiation therapy or IMRT.

ELIGIBILITY:
Inclusion Criteria:

* endometrial adenocarcinoma histologically proven
* post op pelvic radiotherapy
* age ≥ 70
* performance status ≤ 2
* MMSE ≥ 10
* life expectancy ≥ 3 months
* social security covered
* signed informed consent

Exclusion Criteria:

* type I stade IAGI and stade IAGIII without myometer infiltration, stade IIIc2 and IV adenocarcinoma
* uterine sarcoma
* surgery not in accordance with recommendations of Inca
* previous uncontrolled or less than 5 years prior to diagnosis cancer
* cons-indication for radiotherapy
* diarrhea ≥ 3 per day
* pelvic lymph nodes > 1cm not resected during staging
* previous sigmoid diverticulitis, crohn disease, systemic disease, ulcerative haemorrhagic, collagenosis, infectious peritonitis
* IMRT other than tomotherapy
* photon energy < 10MV
* patient under guardianship

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change from baseline in acute toxicity all along the radiation | baseline, Day 5, Day 10, Day 15, Day 20, Day 25, 1 Week after end of treatment, 8 Weeks after end of treatment
  NCI CTCAE v 4.0 tox > grade 2 will be compared

SECONDARY OUTCOMES:
geriatric intervention | up to 6 months
  number of intervention, consequences in terms of base treatment change, intervention of other specialists (except cancer)
geriatric repercussion | baseline, 6 months after end of treatment
  scales : Activities in Daily Living (ADL), Instrumental Activities in Daily Living (IADL), Mini Nutritionnal Assessment (MNA), Geriatric Depression Scale (GDS), cognitive evaluation, Cumulative Illness RAting Scale-Geriatrics (CIRS-G), sociocultural questionnaire, walking and balance
duration of the radiation | up to 5 weeks and a half
  interval between first day and last day of treatment
quality of life | baseline, Day 5, Day 10, Day 15, Day 20, Day 25, 1 week and 8 weeks after end of treatment, 6, 12, 18 and 24 months after end of treatment
  QLQ C30 questionnaire
late major toxicity | 1 week, 8 weeks, 6, 12, 18 and 24 months after the end of treatment
  NCI CTCAE v 4.0
progression free survival | an average period of 2 years
  median time between date of inclusion and date of clinical or radialogical progression

CONTACTS AND LOCATIONS:
Overall Officials: Le Tinier Florence, MD, Principal Investigator — Centre Oscar Lambret
Locations (7):
- France (7):
  - Bergonie Institut, Bordeaux
  - François Baclesse Center, Caen
  - Oscar Lambret Center, Lille
  - Centre Leon Berard, Lyon
  - Institut Jean Godinot, Reims
  - René Gauducheau Center, Saint-Herblain
  - Paul Strauss Center, Strasbourg

IPD SHARING:
Plan to Share IPD: No